CLINICAL TRIAL: NCT06562699
Title: Buffering Capacity of Matcha Green Tea at Two Different Temperatures on Salivary PH After an Acidic Attack: A Randomized Clinical Trial
Brief Title: Buffering Capacity of Matcha Green Tea on Salivary PH After an Acidic Attack
Acronym: ph
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NewGiza University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Allafy, Assistant lecturer, NewGiza University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BC_MGT
Record Dates: First submitted 2024-08-11; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior | interventions — Water

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): 21 participants. They will be generated using numbers from 1 to 63, divided into three groups denoting with letters A, B, and C. Randomization will be generated using (www.randomization.com).
  Interventions: Other: Hot Matcha brew
- Group B (Experimental): 21 participants. They will be generated using numbers from 1 to 63, divided into three groups denoting with letters A, B, and C. Randomization will be generated using (www.randomization.com).
  Interventions: Other: Cold matcha brew
- Group C (Active Comparator): 21 participants. They will be generated using numbers from 1 to 63, divided into three groups denoting with letters A, B, and C. Randomization will be generated using (www.randomization.com).
  Interventions: Other: Water

INTERVENTIONS:
Other: Hot Matcha brew — * Hot matcha brew will be prepared in usucha (thin consistency) version-2 grams of matcha powder (Dr.Baby) mixed with 30 mL of hot water (75 ̊C). The first step will be to massage the matcha powder with a small amount of water until a smooth paste forms, then additional 50 mL of hot water will be added to dilute down the concentration. The matcha will then be vigorously shaken in a lidded jar.
  * After 5 minutes of the acidic attack, participants will be instructed to swish 25 mL of matcha tea 34 times then swallow, and saliva samples will be collected (T2).
  * Then saliva will be collected after 10 (T3), 20 (T4), 30 (T5), and 40 (T6) minutes.
  Arms: Group A
Other: Water — Water (elano) at 13 ̊C swished 34 times then swallowed.
  Arms: Group C
Other: Cold matcha brew — 25 mL of cold matcha brew prepared in usucha (thin consistency) version-2 grams of matcha powder (Dr.Baby) mixed with 80 mL of cold water (13 ̊C) swished 34 times then swallowed.
  Arms: Group B

SUMMARY:
This study is conducted to evaluate the buffering capacity of hot matcha brew in comparison with cold matcha brew and water on salivary pH after an acidic attack using a digital pH meter.

Research Question:

Will matcha green tea beverage have similar salivary buffering effect as water after an acidic challenge on dental interns? Steps in short

1. Recruitment of the patients and clinical examination with medical and dental history taking.
2. Informed consent taking for the eligible participants to participate in the study.
3. A volume of 2 mL saliva samples will be collected before the commencement of acidic attack, baseline (T0).
4. After the acidic attack, saliva will be collected again by spitting method and their pH value will be measured (T1).
5. After 5 minutes of the acidic attack, participants will be instructed to swish either hot matcha tea, cold matcha tea, or water then swallow, and saliva samples will be collected (T2).
6. Then saliva will be collected after 10 (T3), 20 (T4), 30 (T5), and 40 (T6) minutes.

DETAILED DESCRIPTION:
The investigators aim to study the effect of matcha green tea on salivary pH to enhance the volume of scientific awareness and research attention in this area.

Interventions:

Examination:

* For every participant, medical and dental history, caries risk assessment profile, and salivary flow test will be obtained.
* Clinical examination will be done by mouth mirror, explorer, and compressed air through triple syringe to check for active oral diseases.

Trial procedure:

* The participants will be instructed not to brush their teeth in the morning on the day samples will be taken and not to eat or drink until the beginning of the trial to minimize possible food debris and stimulation of saliva.
* The trial time for collecting participants' saliva will be carried out at 09:00-11:00 UTC+2 to prevent any bias in the concentration of saliva due to circadian rhythm.
* Before the beginning of the trial, the pH value of saliva of all participants will be determined. A volume of 2 mL saliva samples will be collected before the commencement of acidic attack, baseline (T0).
* Saliva samples will be collected using spitting method by pooling saliva for 60 s and then spitting in a disposable container sitting in an upright position in a well-lit room with good ventilation. The participants will drool the saliva sample in a 15 mL plastic sterile test tube with lid to prevent CO2 loss to the atmosphere. The salivary sample of each participant will be collected in separate test tubes coded with specific identity number and pH of each sample noted.
* The pH value will be measured with a digital pH meter (AD1030, Adwa Instruments, Hungary) Calibration of the pH meter will be performed before measuring. The glass electrode will be immersed in the saliva sample, and after each measurement, it will be carefully cleaned with deionized water and dried with filter paper. The salivary pH value will be determined by 3 consecutive immersions of the pH meter glass electrode in the test tube with the sample, and the mean value will be taken as the obtained value.
* After the initial salivary pH determination, each participant will be given 25 ml of soft drink (V7 Cola) at room temperature. Participants will be asked to rinse their mouth using 25 ml V7 Cola 34 times and then swallow. Participants will be asked to consume it within 5 minutes of baseline pH.
* Then saliva will be collected again by spitting method and their pH value will be measured (T1).

Intervention:

* Hot matcha brew will be prepared in usucha (thin consistency) version-2 grams of matcha powder (Dr.Baby) mixed with 30 mL of hot water (75 ̊C). The first step will be to massage the matcha powder with a small amount of water until a smooth paste forms, then additional 50 mL of hot water will be added to dilute down the concentration. The matcha will then be vigorously shaken in a lidded jar.
* After 5 minutes of the acidic attack, participants will be instructed to swish 25 mL of matcha tea 34 times then swallow, and saliva samples will be collected (T2).
* Then saliva will be collected after 10 (T3), 20 (T4), 30 (T5), and 40 (T6) minutes.

Comparators:

* First comparator: 25 mL of cold matcha brew prepared in usucha (thin consistency) version-2 grams of matcha powder (Dr.Baby) mixed with 80 mL of cold water (13 ̊C) swished 34 times then swallowed.
* Second comparator: Water (elano) at 13 ̊C swished 34 times then swallowed.

Outcomes Outcomes will be assessed by a digital pH meter (AD1030, Adwa Instruments, Hungary).

Sample size In a previous study by Dehghan et al in 2015 the salivary pH within water group after acidic challenge after 45 minutes was normally distributed with standard deviation 0.56. If the true difference between Matcha green tea and water beverages is 0.5 by using moderate cohen's d effect size, the investigators will need to study 21 patients per group to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05. Sample size was calculated using PS Power and Sample for windows version 3.1.6 using independent t test.

Recruitment Dental interns of New Giza University, Egypt will be recruited for an open-label, parallel group, randomized controlled clinical trial. The selection will be made by the method of random choice. The first 63 interns who register for the offered sessions and meet the criteria for inclusion in the research will be selected as subjects.

Assignment of interventions

Allocation:

Sequence generation H.S. will perform simple randomization according to a check list, including the number of participants by generating numbers from 1 to 63, divided into three groups denoting with letters A, B, and C. Randomization will be generated using (www.randomization.com).

Allocation concealment mechanism The allocation sequence will be kept with H.S. in sealed tight envelopes concealed from the principal investigator A.A. and the outcome assessor E.M. The principal investigator (A.A.) will know the allocation of the consented participant just before starting the trial procedure.

Implementation All participants who fulfill eligibility criteria and who give consent for participation will be randomized by H.S. into three groups.

Blinding (masking):

Outcome assessors will be blinded to the intervention assigned as well as statisticians. Participants cannot be blinded due to the distinctive taste, color, and temperature of different intervention beverages.

Data collection, management, and analysis Data collection methods For every participant, medical and dental history and caries risk assessment profile will be obtained. The examination chart will be filled in by A.A. A.A. will record telephone numbers and addresses of all subjects in the study as a part of the signed consent.

Data management All paper sheets are concerned with the personal or outcome data will be stored in a locked cabinet and in the computer at the Conservative Department. The excel sheets of the patient's data will be stored in the computer of the Conservative Department, School of Dentistry, New Giza University. The computer will have a password known only to A.A. and H.S. to prevent unauthorized access to data and double data entry.

Statistical methods Data will be analyzed using Medcalc software, version 22 for windows (MedCalc Software Ltd, Ostend, Belgium). Continuous data will be described using mean and standard deviation. Intergroup comparison between continuous variables will be performed using independent t test and intragroup comparison will be done using repeated measures ANOVA followed by tukey's post hoc test. A p-value less than or equal to 0.05 will be considered statistically significant and all tests will be two tailed. Statistical power of the study will be set at 80 % with 95 % confidence level.

Monitoring Data monitoring O.M. and H.S. will monitor this study, will have full access to the results, and will take the final decision to terminate the trial.

Harms A.A. should inform participants about possible harms (unpleasant tastes, uncomfortable spitting process). If present, participants should inform the principal investigator and the data will be reported to the main supervisor (H.S.). Harms will be managed through water intake and trial termination.

Auditing In this trial auditing will be done by the main and co-supervisors (O.M. and H.S.) to assure the quality of the research methods and interventions.

ELIGIBILITY:
Inclusion Criteria:

* Low caries-risk.
* Medically healthy.
* Have full permanent dentition.
* Practice daily oral hygiene habits.

Exclusion Criteria:

* Subjects who have active oral diseases as caries, periodontitis, gingivitis, or pulpitis.
* Subjects who have oral-related pain as sensitivity, ulcers, or infection.
* Subjects undergoing restorative or orthodontic treatment.
* Subjects with salivary gland diseases.
* Subjects with systemic diseases.
* Subjects on medications that can affect the salivary gland function (antihistamines, anticancer drugs) in a period of at least two months before the start of the trial.
* Subjects using antibiotics at the time of study or in the period of the last 15 days prior to the study.
* Mouth breathing.
* Smoking.
* Pregnancy.
* Subjects who did not give informed consent.

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Salivary pH buffering effect | 60 minutes
  PH will be assessed by a digital pH meter (AD1030, Adwa Instruments, Hungary). Calibration of the pH meter will be performed before measuring. The glass electrode will be immersed in the saliva sample, and after each measurement, it will be carefully cleaned with deionized water and dried with filter paper. The salivary pH value will be determined by 3 consecutive immersions of the pH meter glass electrode in the test tube with the sample, and the mean value will be taken as the obtained value. Measurements will be taken at baseline, 5 mins after the acidic attack, 5, 10, 20, 30, and 40 minutes after consumption of the buffering beverages.